CLINICAL TRIAL: NCT04726501
Title: A Prospective Multi-center Study for the Treatment of Chinese Children and Adolescents With Newly Diagnosed Hodgkin Lymphoma Using a Modified COG Strategy
Brief Title: CCCG-HD-2018 for Children and Adolescents With Newly Diagnosed Hodgkin Lymphoma
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Children's Cancer Group, China (Network)
Collaborators: Shanghai Children's Medical Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CCCG-HD-2018
Record Dates: First submitted 2021-01-23; First posted 2021-01-27 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Hodgkin Lymphoma
MeSH Terms: conditions — Hodgkin Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Low risk group (Experimental): Ann Arbor stage IA or IIA without bulky disease.
  Interventions: Other: Combined chemotherapy with or without involved-field radiotherapy
- Intermediate risk group (Experimental): Ann Arbor stages IB, IAE, IIB, IIAE, IIIA, IVA with or without bulk disease, and IA or IIA with bulk disease
  Interventions: Other: Combined chemotherapy with or without involved-field radiotherapy
- High risk group (Experimental): Ann Arbor stages III or IV with B symptoms
  Interventions: Other: Combined chemotherapy with or without involved-field radiotherapy

INTERVENTIONS:
Other: Combined chemotherapy with or without involved-field radiotherapy — Patients in low risk group receive 4 cycles of AVE-PC with or without involved-field radiotherapy (IFRT). Patients in intermediate risk group4 cycles ABVE-PC with or without IFRT. RERs in high risk group receive 4 cycles of ABVE-PC followed by followed by IFRT. SERs in high risk group receive 2 cycles of ABVE-PC followed by 2 cycles of IFOS/VINO and 2 cycles of ABVE-PC then followed by IFRT. IFRT consists of 21 Gy in 14 fractions of 1.5 Gy per day and is scheduled within 4 weeks after chemotherapy.

SUMMARY:
The incidence of Hodgkin's lymphoma (HL) in Chinese children and adolescents is only 1 / 10 of that in Europe and the United States, which is a "rare" childhood tumor. Due to the "drug shortage" and extremely low incidence, it has brought great difficulties to the domestic clinical research and failed to achieve the desired effect. In this study, we apply a well-documented effective protocol on newly diagnosed children and adolescents with HL to understand whether the same treatment regimens can obtain similar event free survival rates and overall survival rates and then find out the problems existing in the current clinical care of HL in China, so as to make continuous improvement in the future and prepare for innovative clinical research.

DETAILED DESCRIPTION:
In this study, enrolled patients from age 1 through 18 years with newly diagnosed and biopsy-proven HL are stratified into 3 risk groups according to 3 COG published trials: AHOD0831 (high risk-all Ann Arbor stages III and IV with B symptoms), AHOD0031 (intermediate risk-Ann Arbor stages IB, IAE, IIB, IIAE, IIIA, IVA with or without bulk disease, and IA or IIA with bulk disease) and AHOD0431 (low risk-Ann Arbor stage IA or IIA without bulky disease). Staging was determined with contrast-enhanced CT scanning or MRI, bilateral bone marrow biopsies and FDG-PET. B symptoms included weight loss > 10%, unexplained recurrent fever > 38°, or drenching night sweats. Bulk disease included a mediastinal mass with diameter greater than one third of the thoracic diameter on an upright anterior-posterior (AP) chest radiograph or extramediastinal nodal aggregate > 6 cm in the longest transverse diameter on axial CT.

Low risk group: Patients receive 2 cycles of doxorubicin,vincristine, etoposide, cyclophosphamide, and prednisone (AVE-PC) followed by early response (ER) evaluation. Rapid early responders (RERs) receive 2 additional AVE-PC cycles. Slow early responders (SERs) receive 2 additional ABVE-PC cycles followed by involved-field radiotherapy (IFRT). IFRT consists of 21 Gy in 14 fractions of 1.5 Gy per day and is scheduled within 4 weeks after chemotherapy.

Intermediate risk group: Patients receive 2 cycles of doxorubicin, bleomycin, vincristine, etoposide, cyclophosphamide, and prednisone (ABVE-PC) followed by ER evaluation. RERs receive 2 additional ABVE-PC cycles. SERs receive 2 additional ABVE-PC cycles followed by IFRT. IFRT consists of 21 Gy in 14 fractions of 1.5 Gy per day and is scheduled within 4 weeks after chemotherapy.

High risk group: Patients receive 2 cycles of ABVE-PC followed by ER evaluation. RERs receive 2 additional ABVE-PC cycles followed by IFRT. SERs receive 2 cycles of IFOS/VINO and 2 cycles of ABVE-PC followed by IFRT. IFRT consists of 21 Gy in 14 fractions of 1.5 Gy per day and is scheduled within 4 weeks after chemotherapy.

Patients who have disease progression at any time will be removed from this protocol.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be ages 1 to 18 years at the time of diagnosis; Newly diagnosed, histologically confirmed Hodgkin disease (No nodular lymphocyte-predominant Hodgkin lymphoma)

Exclusion Criteria:

* Patients have received prior cytotoxic chemotherapy for the current diagnosis or any cancer, if any steroid applied, total prior steroids dosage < Prednisone 80 mg/m2; Patients have congenital immunodeficiency, HIV infection, or prior organ transplant; Patients have overwhelming infection, and a life expectancy of < 2 weeks

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 200 (Estimated)
Dates: Start 2018-04-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Event free survival (EFS) | 5 year EFS
  EFS was measured from the day of diagnosis to an event (relapse or progression, death for any reason, abandonment of treatment, second malignancy) or to the date of the last follow-up contact.

SECONDARY OUTCOMES:
Overall survival (OS) | 5 year OS
  OS was measured from the day of diagnosis to the date of death.

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - West China Second University Hospital, Sichuan University, Chengdu, China, Chengdu
  - Nanjing Children's Hospital of Nanjing Medical University, Nanjing, Jiangsu, China, Nanjing
  - Shanghai Children's Medical Center, Shanghai

IPD SHARING:
Plan to Share IPD: Yes
Each centre was responsible for its own data collection. A predefined set of data was collected on protocol-specific forms for each patient and sent to a coordinating center where the findings were reviewed for consistency and completeness. The data were transferred every 12 months. All 12-month reports were reviewed by each local investigator.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: The data were transferred every 12 months during the study period.
Access Criteria: All the data is sharing through paper work every 12 months and meeting discussion every year.

REFERENCES:
- [Background] Kahn JM, Kelly KM, Pei Q, Bush R, Friedman DL, Keller FG, Bhatia S, Henderson TO, Schwartz CL, Castellino SM. Survival by Race and Ethnicity in Pediatric and Adolescent Patients With Hodgkin Lymphoma: A Children's Oncology Group Study. J Clin Oncol. 2019 Nov 10;37(32):3009-3017. doi: 10.1200/JCO.19.00812. Epub 2019 Sep 20. PMID 31539308
- [Background] Friedman DL, Chen L, Wolden S, Buxton A, McCarten K, FitzGerald TJ, Kessel S, De Alarcon PA, Chen AR, Kobrinsky N, Ehrlich P, Hutchison RE, Constine LS, Schwartz CL. Dose-intensive response-based chemotherapy and radiation therapy for children and adolescents with newly diagnosed intermediate-risk hodgkin lymphoma: a report from the Children's Oncology Group Study AHOD0031. J Clin Oncol. 2014 Nov 10;32(32):3651-8. doi: 10.1200/JCO.2013.52.5410. Epub 2014 Oct 13. PMID 25311218
- [Background] Keller FG, Castellino SM, Chen L, Pei Q, Voss SD, McCarten KM, Senn SL, Buxton AB, Bush R, Constine LS, Schwartz CL. Results of the AHOD0431 trial of response adapted therapy and a salvage strategy for limited stage, classical Hodgkin lymphoma: A report from the Children's Oncology Group. Cancer. 2018 Aug 1;124(15):3210-3219. doi: 10.1002/cncr.31519. Epub 2018 May 8. PMID 29738613
- [Background] Gao YJ, Tang JY, Pan C, Lu FJ, Xue HL, Chen J. Risk-adapted chemotherapy without procarbazine in treatment of children with Hodgkin lymphoma. World J Pediatr. 2013 Feb;9(1):32-5. doi: 10.1007/s12519-012-0390-0. Epub 2012 Dec 29. PMID 23275102